CLINICAL TRIAL: NCT03524508
Title: Randomized Phase II Trial of Fluorouracil and Folinic Acid With or Without Liposomal Irinotecan (ONIVYDE) for Patients With Metastatic Biliary Tract Cancer Which Progressed Following Gemcitabine Plus Cisplatin
Brief Title: Nal-IRI(Nanoliposomal Irinotecan) Plus 5-FU/LV in Metastatic Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changhoon Yoo (Other)
Collaborators: Ulsan University Hospital (Other); Chungnam National University Hospital (Other); Kyungpook National University Chilgok Hospital (Other); Inje University (Other)
Responsible Party: Sponsor-Investigator, Changhoon Yoo, Assistant Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIFTY
Record Dates: First submitted 2018-04-18; First posted 2018-05-14 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-FU/LV/Onivyde (Experimental): Onivyde 70 mg/m2 (90 minutes), dl-LV 400mg/m2 or l-LV 200mg/m2 (30 minutes), 5-FU 2400 mg/m2 (46 hours) IV every 2 weeks.
  Interventions: Drug: Onivyde; Drug: 5-FU/LV
- 5FU/LV (Active Comparator): dl-LV 400mg/m2 or l-LV 200mg/m2 (30 minutes), 5-FU 2400 mg/m2 (46 hours) IV every 2 weeks.
  Interventions: Drug: 5-FU/LV

INTERVENTIONS:
Drug: Onivyde — The recommended dose and regimen of Onivyde is 70 mg/m2 intravenously over 90 minutes, followed by dl-LV 400mg/m2 or l-LV 200mg/m2 intravenously over 30 minutes, followed by 5-FU 2400 mg/m2 intravenously over 46 hours, administered every 2 weeks.
  Other Names: Liposomal irinotecan
  Arms: 5-FU/LV/Onivyde
Drug: 5-FU/LV — The recommended dose and regimen of dl-LV 400mg/m2 or l-LV 200mg/m2 intravenously over 30 minutes, followed by 5-FU 2400 mg/m2 intravenously over 46 hours, administered every 2 weeks
  Other Names: Fluorouracil/Folinic acid

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of combination of fluorouracil/folinic acid and liposomal irinotecan(Onivyde) compared with fluoruracil/folinic acid in patients with metastatic biliary tract cancer which progressed on 1st line gemcitabine/cisplatin.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, randomized, phase II study comparing the efficacy and safety between fluorouracil/folinic acid plus liposomal irinotecan and fluoruracil/folinic acid monotherapy in patients with metastatic biliary tract cancer which progressed on 1st line gemcitabine/cisplatin.

Eligible patients will be included in this study and treated according to the protocol. Study treatment will be continued until disease progression, unacceptable toxicity, or patient's decision/consent withdrawal. Local investigators will determine disease progression, radiologic or clinical deterioration.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and written informed consent form
2. ≥ 19 years of age
3. Histologically or cytologically confirmed cholangiocarcinoma
4. Documented metastatic disease
5. At least one measurable lesion according to the RECIST v1.1
6. Disease progression on gemcitabine-cisplatin combination therapy
7. For patients whose disease recurred after curative resection (R0 or R1), previous adjuvant 5-FU-based chemotherapy is allowed if there is at least 6 month-interval between the last dose of adjuvant chemotherapy and recurrence of disease.
8. Adequate hepatic, renal and hematological function AST(Aspartate Aminotransferase), ALT(Alanine Aminotransferase) ≤ 100 IU/L (100 U/L), Cr(Creatinine) ≤ 1.5mg/dL
9. Eastern Cooperative Oncology Group (ECOG) Performance status 0-1

Exclusion Criteria:

1. Serum total bilirubin ≥2 x ULN(upper limit of normal) (biliary drainage is allowed for biliary obstruction)
2. Severe renal impairment (Clcr ≤ 30 ml/min)
3. Inadequate bone marrow reserves as evidenced by:

   * ANC(Absolute Neutrophile Count) ≤ 1,500 cells/μl; or
   * Platelet count ≤ 100,000 cells/μl; or
   * Hemoglobin ≤ 9 g/dL
4. ECOG performance status 2-4
5. Any clinically significant disorder impacting the risk-benefit balance negatively per physician's judgment
6. Any clinically significant gastrointestinal disorder, including hepatic disorders, bleeding, inflammation, occlusion, or diarrhea > grade 2
7. Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) in last 6 months
8. NYHA(New York Heart Association) Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure. Or known abnormal ECG with clinically significant abnormal findings
9. Active infection or an unexplained fever >38.5°C (excluding tumor fever), which in the physician's opinion might compromise the patient's health
10. Current use or any use in last two weeks of strong CYP3A-enzyme inducers/inhibitors and/or strong UGT1A inhibitors
11. Known hypersensitivity to any of the components of Onivyde other liposomal irinotecan formulations, irinotecan, fluoropyrimidines, or leucovorin.
12. Breast feeding, known pregnancy, positive serum pregnancy test or unwillingness to use an effective method of contraception, during therapy and for 3 months following the last dose of Onivyde. Females of Childbearing Potential must either agree to use and be able to take effective contraceptive birth control measures (Pearl Index < 1) or agree to practice complete abstinence from heterosexual intercourse during the course of the study and for at least 3 months after last application of program treatment. A female subject is considered to be of childbearing potential unless she is age ≥ 50 years and naturally amenorrhoeic for ≥ 2 years, or unless she is surgically sterile. Males must agree not to father a child (including not donating sperm) during the course of the trial and for at least 6 months after last administration of study drugs.
13. Previous treatment with combination drug tegafur, gimeracil, and oteracil potassium with seven days before enrollment.
14. Current treatment with Sorivudine.
15. Severe fatigue or bone marrow depression after prior radiotherapy or antineoplastic therapy
16. Pregnancy or women with child-bearing potential or lactating
17. Non-malignant severe co-morbidity
18. Previous second-line anti-cancer therapy (e.g., Tegafur)
19. History of other malignancy with a disease-free interval <5 years (Registration is permitted if it has minimal impact on prognosis, such as carcinoma in situ and papillary thyroid cancer)
20. History or current eveidence of brain metastasis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival by independent central reviewer | from the date of enrollment to the earlier of the date of confirmed progression or death from any cause. (assessed up to 36 months)
  Progression-free survival is the time from the date of enrollment to the earlier of the date of confirmed progression or death from any cause.

SECONDARY OUTCOMES:
Overall Survival | from the date of enrollment to death from any cause. (assessed up to 36 months)
  Overall survival is the time from the date of enrollment to death from any cause
Response rates determined by the investigator according to the RECIST(Response Evaluation Criteria in Solid Tumors) v1.1 | from the date of enrollment to end of treatment. (assessed up to 36 months)
  The response rate is the proportion of eligible patients with measurable lesions with a overall response of CR(Complete Response) or PR(Partial Response)
EORTC-QLQ (European Organization for Research and Treatment of Cancer - Quality of life Questionnaire) C30 (version 3.0) | from the date of Screening to end of treatment. (assessed up to 36 months)
  EORTC-QLQ C-30 questionnaires will be performed at screening visit, at pre-dose (Cycle 1 Day1) of every subsequent cycle, at the end of treatment visit. It is a 30-item questionnaire. It has 4-point scales for the item number 1 to 28. These are coded with the same response categories as items 1 to 28, namely "not at all=1" "a little=2" "quite a bit=3" and "very much=4" It has 7-point scale for question number 29 to 30. These are coded with the same response categories as items 29 to 30, namely "worst=1" to "best=7" Total score will be minimum 30 and maximum 126.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | from the date of enrollment to 30 days after last treatment. (assessed up to 36 months)
  Severity of adverse events will be graded by NCI-CTCAE (National Cancer Institute - Common Terminology Criteria for Adverse Events) v4.03
Progression Free Survival by investigator assessment | from the date of enrollment to the earlier of the date of confirmed progression or death from any cause. (assessed up to 36 months)
  Progression-free survival is the time from the date of enrollment to the earlier of the date of confirmed progression or death from any cause.
Response rates determined by the independent central reviewer | from the date of enrollment to end of treatment. (assessed up to 36 months)
  The response rate is the proportion of eligible patients with measurable lesions with a overall response of CR(Complete Response) or PR(Partial Response)

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Edge SB, Compton CC. The American Joint Committee on Cancer: the 7th edition of the AJCC cancer staging manual and the future of TNM. Ann Surg Oncol. 2010 Jun;17(6):1471-4. doi: 10.1245/s10434-010-0985-4. PMID 20180029
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Okusaka T, Nakachi K, Fukutomi A, Mizuno N, Ohkawa S, Funakoshi A, Nagino M, Kondo S, Nagaoka S, Funai J, Koshiji M, Nambu Y, Furuse J, Miyazaki M, Nimura Y. Gemcitabine alone or in combination with cisplatin in patients with biliary tract cancer: a comparative multicentre study in Japan. Br J Cancer. 2010 Aug 10;103(4):469-74. doi: 10.1038/sj.bjc.6605779. Epub 2010 Jul 13. PMID 20628385
- [Background] Valle JW, Borbath I, Khan SA, Huguet F, Gruenberger T, Arnold D; ESMO Guidelines Committee. Biliary cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2016 Sep;27(suppl 5):v28-v37. doi: 10.1093/annonc/mdw324. No abstract available. PMID 27664259
- [Background] Kim BJ, Hyung J, Yoo C, Kim KP, Park SJ, Lee SS, Park DH, Song TJ, Seo DW, Lee SK, Kim MH, Park JH, Cho H, Ryoo BY, Chang HM. Prognostic factors in patients with advanced biliary tract cancer treated with first-line gemcitabine plus cisplatin: retrospective analysis of 740 patients. Cancer Chemother Pharmacol. 2017 Jul;80(1):209-215. doi: 10.1007/s00280-017-3353-2. Epub 2017 Jun 8. PMID 28597043
- [Background] Fornaro L, Cereda S, Aprile G, Di Girolamo S, Santini D, Silvestris N, Lonardi S, Leone F, Milella M, Vivaldi C, Belli C, Bergamo F, Lutrino SE, Filippi R, Russano M, Vaccaro V, Brunetti AE, Rotella V, Falcone A, Barbera MA, Corbelli J, Fasola G, Aglietta M, Zagonel V, Reni M, Vasile E, Brandi G. Multivariate prognostic factors analysis for second-line chemotherapy in advanced biliary tract cancer. Br J Cancer. 2014 Apr 29;110(9):2165-9. doi: 10.1038/bjc.2014.190. Epub 2014 Apr 8. PMID 24714745
- [Background] Lamarca A, Hubner RA, David Ryder W, Valle JW. Second-line chemotherapy in advanced biliary cancer: a systematic review. Ann Oncol. 2014 Dec;25(12):2328-2338. doi: 10.1093/annonc/mdu162. Epub 2014 Apr 25. PMID 24769639
- [Background] Brieau B, Dahan L, De Rycke Y, Boussaha T, Vasseur P, Tougeron D, Lecomte T, Coriat R, Bachet JB, Claudez P, Zaanan A, Soibinet P, Desrame J, Thirot-Bidault A, Trouilloud I, Mary F, Marthey L, Taieb J, Cacheux W, Lievre A. Second-line chemotherapy for advanced biliary tract cancer after failure of the gemcitabine-platinum combination: A large multicenter study by the Association des Gastro-Enterologues Oncologues. Cancer. 2015 Sep 15;121(18):3290-7. doi: 10.1002/cncr.29471. Epub 2015 Jun 5. PMID 26052689
- [Background] Kim BJ, Yoo C, Kim KP, Hyung J, Park SJ, Ryoo BY, Chang HM. Efficacy of fluoropyrimidine-based chemotherapy in patients with advanced biliary tract cancer after failure of gemcitabine plus cisplatin: retrospective analysis of 321 patients. Br J Cancer. 2017 Feb 28;116(5):561-567. doi: 10.1038/bjc.2016.446. Epub 2017 Jan 12. PMID 28081540
- [Background] Innocenti F, Kroetz DL, Schuetz E, Dolan ME, Ramirez J, Relling M, Chen P, Das S, Rosner GL, Ratain MJ. Comprehensive pharmacogenetic analysis of irinotecan neutropenia and pharmacokinetics. J Clin Oncol. 2009 Jun 1;27(16):2604-14. doi: 10.1200/JCO.2008.20.6300. Epub 2009 Apr 6. PMID 19349540
- [Background] Bellanti F, Kagedal B, Della Pasqua O. Do pharmacokinetic polymorphisms explain treatment failure in high-risk patients with neuroblastoma? Eur J Clin Pharmacol. 2011 May;67 Suppl 1(Suppl 1):87-107. doi: 10.1007/s00228-010-0966-3. Epub 2011 Feb 2. PMID 21287160
- [Background] Mathijssen RH, van Alphen RJ, Verweij J, Loos WJ, Nooter K, Stoter G, Sparreboom A. Clinical pharmacokinetics and metabolism of irinotecan (CPT-11). Clin Cancer Res. 2001 Aug;7(8):2182-94. PMID 11489791
- [Background] Kawato Y, Aonuma M, Hirota Y, Kuga H, Sato K. Intracellular roles of SN-38, a metabolite of the camptothecin derivative CPT-11, in the antitumor effect of CPT-11. Cancer Res. 1991 Aug 15;51(16):4187-91. PMID 1651156
- [Background] Garcia-Carbonero R, Supko JG. Current perspectives on the clinical experience, pharmacology, and continued development of the camptothecins. Clin Cancer Res. 2002 Mar;8(3):641-61. PMID 11895891
- [Background] Vanhoefer U, Harstrick A, Achterrath W, Cao S, Seeber S, Rustum YM. Irinotecan in the treatment of colorectal cancer: clinical overview. J Clin Oncol. 2001 Mar 1;19(5):1501-18. doi: 10.1200/JCO.2001.19.5.1501. PMID 11230497
- [Background] Drummond DC, Noble CO, Guo Z, Hong K, Park JW, Kirpotin DB. Development of a highly active nanoliposomal irinotecan using a novel intraliposomal stabilization strategy. Cancer Res. 2006 Mar 15;66(6):3271-7. doi: 10.1158/0008-5472.CAN-05-4007. PMID 16540680
- [Background] Kang MH, Wang J, Makena MR, Lee JS, Paz N, Hall CP, Song MM, Calderon RI, Cruz RE, Hindle A, Ko W, Fitzgerald JB, Drummond DC, Triche TJ, Reynolds CP. Activity of MM-398, nanoliposomal irinotecan (nal-IRI), in Ewing's family tumor xenografts is associated with high exposure of tumor to drug and high SLFN11 expression. Clin Cancer Res. 2015 Mar 1;21(5):1139-50. doi: 10.1158/1078-0432.CCR-14-1882. PMID 25733708
- [Background] Kalra AV, Kim J, Klinz SG, Paz N, Cain J, Drummond DC, Nielsen UB, Fitzgerald JB. Preclinical activity of nanoliposomal irinotecan is governed by tumor deposition and intratumor prodrug conversion. Cancer Res. 2014 Dec 1;74(23):7003-13. doi: 10.1158/0008-5472.CAN-14-0572. Epub 2014 Oct 1. PMID 25273092
- [Background] Tsai CS, Park JW, Chen LT. Nanovector-based therapies in advanced pancreatic cancer. J Gastrointest Oncol. 2011 Sep;2(3):185-94. doi: 10.3978/j.issn.2078-6891.2011.034. PMID 22811849
- [Background] Benson AB 3rd, Ajani JA, Catalano RB, Engelking C, Kornblau SM, Martenson JA Jr, McCallum R, Mitchell EP, O'Dorisio TM, Vokes EE, Wadler S. Recommended guidelines for the treatment of cancer treatment-induced diarrhea. J Clin Oncol. 2004 Jul 15;22(14):2918-26. doi: 10.1200/JCO.2004.04.132. PMID 15254061
- [Background] Wang-Gillam A, Li CP, Bodoky G, Dean A, Shan YS, Jameson G, Macarulla T, Lee KH, Cunningham D, Blanc JF, Hubner RA, Chiu CF, Schwartsmann G, Siveke JT, Braiteh F, Moyo V, Belanger B, Dhindsa N, Bayever E, Von Hoff DD, Chen LT; NAPOLI-1 Study Group. Nanoliposomal irinotecan with fluorouracil and folinic acid in metastatic pancreatic cancer after previous gemcitabine-based therapy (NAPOLI-1): a global, randomised, open-label, phase 3 trial. Lancet. 2016 Feb 6;387(10018):545-557. doi: 10.1016/S0140-6736(15)00986-1. Epub 2015 Nov 29. PMID 26615328
- [Derived] Yoo C, Saborowski A, Hyung J, Wenzel P, Kim I, Wege H, Kim KP, Folprecht G, Ryoo BY, Schutt P, Cheon J, Gotze T, Ryu H, Lee JS, Vogel A. Liposomal irinotecan for previously treated patients with biliary tract cancer: A pooled analysis of NIFTY and NALIRICC trials. J Hepatol. 2025 Oct;83(4):909-916. doi: 10.1016/j.jhep.2025.03.013. Epub 2025 Mar 25. PMID 40147791
- [Derived] Hyung J, Kim I, Kim KP, Ryoo BY, Jeong JH, Kang MJ, Cheon J, Kang BW, Ryu H, Lee JS, Kim KW, Abou-Alfa GK, Yoo C. Treatment With Liposomal Irinotecan Plus Fluorouracil and Leucovorin for Patients With Previously Treated Metastatic Biliary Tract Cancer: The Phase 2b NIFTY Randomized Clinical Trial. JAMA Oncol. 2023 May 1;9(5):692-699. doi: 10.1001/jamaoncol.2023.0016. PMID 36951834
- [Derived] Yoo C, Kim KP, Jeong JH, Kim I, Kang MJ, Cheon J, Kang BW, Ryu H, Lee JS, Kim KW, Abou-Alfa GK, Ryoo BY. Liposomal irinotecan plus fluorouracil and leucovorin versus fluorouracil and leucovorin for metastatic biliary tract cancer after progression on gemcitabine plus cisplatin (NIFTY): a multicentre, open-label, randomised, phase 2b study. Lancet Oncol. 2021 Nov;22(11):1560-1572. doi: 10.1016/S1470-2045(21)00486-1. Epub 2021 Oct 14. PMID 34656226
- See also: Camptosar® (irinotecan) U.S. Package Insert (Accessed 23 March 2016) — http://www.accessdata.fda.gov/drugsatfda_docs/label/2014/020571s048lbl.pdf
- See also: Irinotecan hydrochloride Summary of Product Characteristics (Accessed 23 March 2016) — https://www.medicines.org.uk/emc/medicine/21586